CLINICAL TRIAL: NCT05626413
Title: Cardiovascular Disease and Diabetes in Silesian Patients
Brief Title: Cardiovascular Disease in Patients With Diabetes: The Silesia Diabetes-Heart Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Collaborators: Silesian University of Technology (Other); Liverpool Centre for Cardiovascular Science at University of Liverpool, Liverpool John Moores University and Liverpool Heart & Chest Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Silesia Diabetes-Heart Project
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
Keywords: Cardiovascular disease; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project is an observational one which undertakes different, easy to obtain in everyday clinical practice, demographical, laboratory and clinical parameters of patients with diabetes in Silesian Region in Poland to predict cardiovascular disease, cardiovascular events and neuropathy using machine learning approach.

DETAILED DESCRIPTION:
The study is a prospective, observational one in which it is planned to obtain demographical, laboratory and clinical parameters of patients who are hospitalized in one the the main diabetology sites in Silesia region in Poland and to follow them prospectively for 10 years in order to collect information related to new cardiovascular events. Telephone contact will be performed every 12 months following hospital discharge. Any procedures related to the patients hospitalized in the diabetology ward will be the routine ones and the bioethics committee of Medical University of Silesia gave the permission for the study but waved the necessity of informed consent to be signed.Moreover there will be subgroup analysis of patients recruited from the outpatient diabetology clinics in Silesia region in order to participate in the observational study collecting data related to to vitamin D concentration, densitometry, fibroscan, carotid ultrasound examination, vascular stiffness, electrocardiography, peripheral and cardiovascular autonomic neuropathy and fundus imaging. Patients who are treated in outpatient diabetology clinics in Silesia region and are included into the study must have the informed consent signed and bioethics committee agreement has been obtained.

Machine learning approach will be implemented to discover the association between easy to obtain in everyday practice parameters, namely clinical, biochemical, and demographical ones to identify patients at the highest risk of cardiovascular disease.

The secondary aim of the study is to utilize fundus imaging, electrocardiography, alongside demographic and clinical data in order to potentially diagnose neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* For the group of hospitalized patients: diabetes type 1 or type 2
* For the subgroup of patients treated in outpatient diabetology clinics in Silesia region: diabetes type 1 or type 2

Exclusion Criteria:

1. For the group of hospitalized patients:

   * Types of diabetes other than type 1 and type 2 diabetes
   * Death during hospital stay
   * Terminal stage of cancer.
2. For the subgroup of patients recruited form outpatient diabetology clinics:

   * Lack of an informed consent
   * Types of diabetes other than type 1 and type 2 diabetes
   * Malignant neoplasms
   * Terminal stage of neoplasm
   * End-stage renal disease
   * Malabsorption syndrome
   * Active infection
   * Primary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in diabetology ward in Zabrze. Patients treated in outpatient diabetology clinics in Silesia region.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The risk of cardiovascular disease and events among patients with diabetes | 5 years
  To predict the risk of cardiovascular disease and events among patients with diabetes using machine learning approach

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Nabrdalik, PhD,prof., Principal Investigator — Medical University of Silesia
Locations (1):
- Department of Internal Diseases, Diabetology and Nephrology, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janota O, Mantovani M, Kwiendacz H, Irlik K, Bucci T, Lam SHM, Huang B, Alam U, Boriani G, Hendel M, Piasnik J, Olejarz A, Wlosowicz A, Pabis P, Wojcik W, Gumprecht J, Lip GYH, Nabrdalik K. Metabolically "extremely unhealthy" obese and non-obese people with diabetes and the risk of cardiovascular adverse events: the Silesia Diabetes - Heart Project. Cardiovasc Diabetol. 2024 Sep 3;23(1):326. doi: 10.1186/s12933-024-02420-x. PMID 39227929
- [Derived] Nabrdalik K, Irlik K, Meng Y, Kwiendacz H, Piasnik J, Hendel M, Ignacy P, Kulpa J, Kegler K, Herba M, Boczek S, Hashim EB, Gao Z, Gumprecht J, Zheng Y, Lip GYH, Alam U. Artificial intelligence-based classification of cardiac autonomic neuropathy from retinal fundus images in patients with diabetes: The Silesia Diabetes Heart Study. Cardiovasc Diabetol. 2024 Aug 10;23(1):296. doi: 10.1186/s12933-024-02367-z. PMID 39127709
- [Derived] Nabrdalik K, Kwiendacz H, Irlik K, Hendel M, Drozdz K, Wijata AM, Nalepa J, Janota O, Wojcik W, Gumprecht J, Lip GYH. Machine learning identification of risk factors for heart failure in patients with diabetes mellitus with metabolic dysfunction associated steatotic liver disease (MASLD): the Silesia Diabetes-Heart Project. Cardiovasc Diabetol. 2023 Nov 20;22(1):318. doi: 10.1186/s12933-023-02014-z. PMID 37985994